CLINICAL TRIAL: NCT07195318
Title: Low-dose Fisetin Supplementation for Healthy Aging - a Triple-blind, Randomized, Placebo-controlled Trial
Brief Title: Fisetin Supplementation for Healthy Aging
Acronym: Fisetin LOW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ove Andersen (Other)
Responsible Party: Sponsor-Investigator, Ove Andersen, Head of Research, Clinical Professor, Principal Investigator, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-25043857
Record Dates: First submitted 2025-09-12; First posted 2025-09-26 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Chronic inflammation; Cellular senescence; Senotherapeutics
MeSH Terms: interventions — fisetin

STUDY DESIGN:
Intervention Model Description: The study is a 2-arm triple-blind randomized placebo-controlled trial, in which middle-aged and older adults will receive either:
  * 100 mg fisetin daily for 7 weeks (intervention group), or
  * placebo daily for 7 weeks (control group).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Fisetin daily for 7 weeks
  Interventions: Dietary Supplement: Fisetin
- Placebo group (Placebo Comparator): Placebo daily for 7 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fisetin — One capsule (100 mg) daily
  Arms: Treatment group
Dietary Supplement: Placebo — One capsule daily
  Arms: Placebo group

SUMMARY:
There is growing interest among the general population in preventive health interventions that can help mitigate age-related decline, reduce the risk of chronic diseases, and promote healthy aging. The use of nutritional supplements has been increasing and is especially high in older adults and healthier individuals. In response to this demand, a growing number of nutritional supplements are being advertised for their "anti-aging" properties, claiming to target molecular and cellular "hallmarks of aging", such as chronic inflammation, oxidative stress, and cellular senescence. However, the overwhelming majority of these claims stem from preclinical studies in animal models (e.g., C. elegans, mice), and there is extremely limited evidence for beneficial effects, effective doses, or safety profiles of these supplements in humans. Moreover, the lack of strict regulations in the nutritional supplement industry leads to wide differences in the quality and in the actual content of active substances between supplements, which could impact both their efficacy and safety.

The investigators will conduct a clinical trial in healthy volunteers, who will receive supplementation with fisetin (100 mg) or placebo daily for 7 weeks. Participants will be examined at regular intervals during the study period. The investigators will then investigate whether fisetin supplementation is safe and evaluate its effect on measures of chronic inflammation, cellular senescence, aging, and general health.

DETAILED DESCRIPTION:
The goal of this study is to assess the anti-inflammatory effects, overall health benefits, and the safety of a daily low dose (100 mg) of fisetin in relatively healthy middle-aged and older adults.

The study is a 2-arm triple-blind randomized placebo-controlled trial, in which middle-aged and older adults (n=120) will receive either:

* One capsule (100 mg) fisetin daily for 7 weeks (intervention group), or
* One capsule placebo daily for 7 weeks (control group).

ELIGIBILITY:
Inclusion Criteria:

* Middle-aged or older adult (≥50 years),
* Able to cooperate cognitively,
* Able to read and understand Danish,

Exclusion Criteria:

* Inability or unwillingness to take oral supplements,
* Chronic or recent (within 30 days) use of other anti-aging supplements,
* Chronic or recent (within 30 days) treatment with medications having anti-aging effects (e.g., metformin, rapamycin, semaglutide),
* Chronic or recent (within 30 days) treatment with anti-inflammatory medications,
* Chronic or recent (within 30 days) treatment with the medications that can interact negatively with fisetin,
* Recent (within 14 days) vaccination,
* Treatment with another investigational drug or other intervention within 1 year,
* Active cancer or current cancer treatment,
* Unstable or uncontrolled major disorders, e.g., cardiovascular, renal, endocrine, immunological, hepatic disorder, or cancer, requiring regular monitoring at the hospital
* Planned medical and surgical procedures during the study period,
* Known hypersensitivity or allergy to fisetin or excipients in the placebo capsules,
* Presence of any condition that the investigator believes would put the participant at risk or would preclude the participant from successfully completing all aspects of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2035-09-20 (Estimated)

PRIMARY OUTCOMES:
Soluble urokinase plasminogen activator receptor (suPAR) | Baseline to Week 7
  The difference between groups in the change in plasma levels of suPAR

SECONDARY OUTCOMES:
Side effects | Baseline to Week 7
  Differences between groups in the type and frequency of side effects

OTHER OUTCOMES:
SASP factors and inflammation markers | Baseline to Week 7
  Differences between groups in the change in plasma concentrations (pg/mL) of SASP factors and inflammation markers (e.g., cytokines, chemokines, proteases, growth factors).
Cellular senescence | Baseline to Week 7
  Differences between groups in the change in the percentage of immune cells positive for expression of senescence markers (e.g., p16INK4a, p21CIP1/WAF1, SA-B-gal) .
Aging biomarkers | Baseline to Week 7
  Differences between groups in the change in plasma concentrations (pg/mL) of aging markers (e.g., α-klotho, growth differentiation factor 15, fibroblast growth factor 21).
Frailty | Baseline to Week 7
  Differences between groups in the change in frailty status calculated as Frailty Index OutRef (FI-OutRef) based on the values of 17 routine biochemistry biomarkers. The score ranges from 0-17, with higher scores indicating greater frailty.
Clinical biomarkers | Baseline to Week 7
  Differences between groups in the change in levels of routine biochemistry markers (e.g., alanine aminotransferase, albumin, alkaline phosphatase, bilirubin, blood urea nitrogen, coagulation factors II, VII and X, CRP, creatinine, hemoglobin, lactate dehydrogenase, mean corpuscular hemoglobin concentration, mean corpuscular volume, neutrophils, potassium, sodium, thrombocytes, white blood cell count, cystatin C, cholesterol (total, low-density lipoproteins, high-density lipoproteins), triglycerides, and hemoglobin A1c).
Physical function | Baseline to Week 7
  Differences between groups in the change in gait speed (m/s).
Physical function | Baseline to Week 7
  Differences between groups in the change in hand grip strength (kg).
Physical function | Baseline to Week 7
  Differences between groups in the change in chair stand test score (number of repetitions).
Physical function | Baseline to Week 7
  Differences between groups in the change in balance score (0-4 points, with higher scores indicating poorer balance).
Cognitive function | Baseline to Week 7
  Differences between groups in the change in cognitive function assessed using the Montreal Cognitive Assessment (MoCA) score (0-30, with higher values indicating better cognitive function).
Cognitive function | Baseline to Week 7
  Differences between groups in the change in cognitive function assessed using the Digit Symbol Substitution Test (DSST), with higher scores indicating better cognitive function.
Health-related quality of life | Baseline to Week 7
  Differences between groups in the change in quality of life assessed using the EuroQol-5D-5L. The score ranges from 1 to -0.757, which higher values indicating better quality of life.
Self-rated health | Baseline to Week 7
  Differences between groups in the change in self-rated health, classified as excellent, very good, good, fair, or poor.
CYP3A4 activity | Baseline to Week 7
  Differences between groups in the change in CYP3A4 activity assessed using the concentration of the endogenous marker 4β-hydroxycholesterol measured in plasma samples using LC-MS/MS.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette Tavenier, Study Chair — Copenhagen University Hospital, Amager and Hvidovre; Line Jee Hartmann Rasmussen, Study Chair — Copenhagen University Hospital, Amager and Hvidovre; Morten B Houlind, Study Chair — Copenhagen University Hospital, Amager and Hvidovre; Magnus Berglind, Study Chair — Copenhagen University Hospital, Amager and Hvidovre; Line Fleischer Hach, Study Chair — Copenhagen University Hospital, Amager and Hvidovre
Locations (1):
- Department of Clinical Research, Copenhagen University Hospital Amager & Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided